CLINICAL TRIAL: NCT00498992
Title: Regenecare® in the Treatment of Skin Rash Associated With Cetuximab (Erbitux®) or Other EGFR Treated Cancer Patients
Brief Title: Regenecare® Wound Gel in Treating Rash in Patients Receiving Cetuximab or Other Epidermal Growth Factor Receptor Inhibitor Therapy for Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ingalls Memorial Hospital (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: CDR0000553120; IMH-REG-ING-100; MPMM-IMH-REG-ING-100
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-07

CONDITIONS: Dermatologic Complications; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: dermatologic complications; unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Dietary Supplement: collagen/aloe vera/vitamin E/lidocaine topical hydrogel

SUMMARY:
RATIONALE: Regenecare® wound gel may help relieve pain and itching in patients who develop an acne-like rash while undergoing treatment with cetuximab or another epidermal growth factor receptor inhibitor for cancer.

PURPOSE: This clinical trial is studying how well Regenecare® wound gel works in treating rash in patients receiving cetuximab or another epidermal growth factor receptor inhibitor therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of Regenecare® wound gel in alleviating pain and itching in patients who develop an acneiform rash while undergoing treatment with cetuximab or other EGFR inhibitor therapy for cancer.

Secondary

* Determine the efficacy of this drug in reducing the severity of rash in these patients.
* Determine the efficacy of this drug in reducing the redness and appearance of the rash in these patients.
* Determine the tolerability of this drug in these patients.

OUTLINE: This is a prospective study.

* Observation: Patients undergo evaluation by full-face photography prior to development of skin rash (baseline). While undergoing concurrent cancer therapy, patients self-monitor for the appearance of an acneiform rash. Upon initial onset of rash, patients proceed to treatment.
* Treatment: Patients apply topical Regenecare® wound gel to the face ≥ 4 times daily. Treatment continues for 4 weeks in the absence of unacceptable toxicity.

Patients are evaluated weekly by facial examination, full-face photography, and patient satisfaction questionnaires.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Starting treatment with cetuximab or other EGFR inhibitor (e.g., erlotinib hydrochloride) on another clinical trial

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* No known history of hypersensitivity to amine-type local anesthetics or to other components of MPM Regenecare® wound gel
* No other concurrent, serious skin disorders (i.e., scleroderma or psoriasis) that would interfere with assessment of EGFR inhibitor-induced rash

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No other concurrent topical facial creams or lotions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-07

PRIMARY OUTCOMES:
Efficacy of Regenecare® wound gel, in terms of alleviating pain and itching

SECONDARY OUTCOMES:
Efficacy of Regenecare® wound gel, in terms of reducing severity, redness, and appearance of rash
Tolerability of Regenecare® wound gel as assessed by NCI CTCAE v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Mark F. Kozloff, MD, Study Chair — Ingalls Memorial Hospital
Locations (1):
- Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois, United States